CLINICAL TRIAL: NCT07380529
Title: Comparison of the Effect of Carbetocin Versus Oxytocin in the Prevention of Postpartum Hemorrhage After Emergency Caesarean Section in Antenatal Low-risk Patients
Acronym: EMERGE-CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Tahir Eryılmaz, Gynecology and Obstetrics M.D. specialist, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AEŞH-EKI-2024-0025
Record Dates: First submitted 2026-01-18; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Hemorrhage (PPH)
Keywords: carbetocin; postpartum hemorrhage; oxytocin; emergency caesarean delivery
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Oxytocin (Active Comparator): Standard oxytocin regimen after delivery (uterotonic prophylaxis at emergency cesarean)
  Interventions: Drug: Oxytocin
- carbetocin (Experimental): Carbetocin administered as a single dose immediately after delivery during emergency cesarean section for prophylaxis of postpartum hemorrhage
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — Carbetocin administered as a single dose immediately after delivery during emergency cesarean section for prophylaxis of postpartum hemorrhage
  Arms: carbetocin
Drug: Oxytocin — Oxytocin administered per institutional standard regimen immediately after delivery during emergency cesarean section for prophylaxis of postpartum hemorrhage
  Arms: Oxytocin

SUMMARY:
This study will be conducted to compare the effects of pabal and oxytocin administered to prevent postpartum hemorrhage in patients who were followed in the delivery room due to vaginal labor but underwent cesarean section due to emergency situations.

DETAILED DESCRIPTION:
The aim of this study is to compare the effectiveness of oxytocin or the long-acting oxytocin analog carbetocin (Pabal) administered to pregnant women to prevent postpartum hemorrhage after emergency cesarean delivery.

The primary aim is to evaluate the amount of postpartum bleeding after the use of these two agents and to identify potential risk factors that may change the effectiveness of these drugs.

The secondary aim is to observe the changes in intraoperative and postoperative hemodynamic parameters after the administration of these two drugs.

According to NICE (National Institute Health and Care) and RCOG (Royal College of Obstetricians and Gynaecologists) guidelines, patients who are in the emergency caesarean category 1 (The life of the mother or baby is in danger. The caesarean should be performed as soon as possible, usually within 30 minutes after the decision is made) group will be included.

The aim of this study is to compare the effectiveness of oxytocin or the long-acting oxytocin analog carbetocin (Pabal) administered to pregnant women to prevent postpartum hemorrhage after emergency cesarean delivery.

The primary aim is to evaluate the amount of postpartum bleeding after the use of these two agents and to identify potential risk factors that may change the effectiveness of these drugs.

The secondary aim is to observe the changes in intraoperative and postoperative hemodynamic parameters after the administration of these two drugs.

According to NICE (National Institute Health and Care) and RCOG (Royal College of Obstetricians and Gynaecologists) guidelines, patients who are in the emergency caesarean category 1 (The life of the mother or baby is in danger. The caesarean should be performed as soon as possible, usually within 30 minutes after the decision is made) group will be included.

The aim of this study is to compare the effectiveness of oxytocin or the long-acting oxytocin analog carbetocin (Pabal) administered to pregnant women to prevent postpartum hemorrhage after emergency cesarean delivery.

The primary aim is to evaluate the amount of postpartum bleeding after the use of these two agents and to identify potential risk factors that may change the effectiveness of these drugs.

The secondary aim is to observe the changes in intraoperative and postoperative hemodynamic parameters after the administration of these two drugs.

According to NICE (National Institute Health and Care) and RCOG (Royal College of Obstetricians and Gynaecologists) guidelines, patients who are in the emergency caesarean category 1 (The life of the mother or baby is in danger. The caesarean should be performed as soon as possible, usually within 30 minutes after the decision is made) group will be included. Patients are routinely informed about the vaginal delivery process when they come into labor. It was planned to inform the women about the medications planned to be given to prevent postpartum hemorrhage in case of a possible emergency caesarean section and to obtain their written consent.

The patient data was designed to be accessible from the hospital information system (Keydata Information Technology Technology Systems), and it was planned to re-check the patient files in order to increase the accuracy and reliability of the data. IBM SPSS Statistics 23.0 (IBM Corp., Armonk, NY, USA) will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria

* Term pregnancy (>37 weeks gestation)
* Singleton pregnancy
* Vertex presentation
* not having had a cesarean section before
* emergency cesarean delivery (category 1)
* low risk for postpartum hemorrhage
* Vaginal labor has started (> 4 cm cervical dilatation) or a decision has been made (rupture of membranes, Abnormal findings on NST or other signs of fetal compromise.) Exclusion Criteria
* Non-term pregnancy (< 37 weeks gestation)
* Non- vertex presentation
* antenatal high risk pregnancy for postpartum hemorrhage (preeclampsia/eclampsia, previous uterine surgery, placental anomalies)
* Twin pregnancy
* Elective cesarean section planned

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Postoperative change in hemoglobin at 24 hours | Baseline (preoperative) and within 24 hours after emergency cesarean delivery
  Change in hemoglobin (g/dL) from preoperative baseline to the lowest hemoglobin value within 24 hours after emergency cesarean delivery, compared between the carbetocin and oxytocin groups.

SECONDARY OUTCOMES:
Need for additional uterotonic agents | Within 24 hours after cesarean delivery
  Proportion of participants requiring any additional uterotonic agent(s) within 24 hours after cesarean delivery (after administration of the assigned study drug).
Postoperative change in hematocrit at 24 hours | Baseline (preoperative) and within 24 hours after emergency cesarean delivery
  Change in hematocrit (%) from preoperative baseline to the lowest hematocrit value within 24 hours after emergency cesarean delivery, compared between the carbetocin and oxytocin groups.

CONTACTS AND LOCATIONS:
Overall Officials: TAHİR ERYILMAZ, M.D. Dr., Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Razali N, Md Latar IL, Chan YK, Omar SZ, Tan PC. Carbetocin compared to oxytocin in emergency cesarean section: a randomized trial. Eur J Obstet Gynecol Reprod Biol. 2016 Mar;198:35-39. doi: 10.1016/j.ejogrb.2015.12.017. Epub 2015 Dec 30. PMID 26773246
- See also: Utilization of carbetocin for prevention of postpartum hemorrhage after cesarean section: a randomized clinical trial — https://link.springer.com/article/10.1007/s00404-009-0973-8